CLINICAL TRIAL: NCT01789788
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO6811135 in Patients With Type 2 Diabetes Mellitus.
Brief Title: A Safety, Pharmacokinetics and Pharmacodynamics Study of RO6811135 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP28436
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO6811135 (Experimental)
  Interventions: Drug: RO6811135

INTERVENTIONS:
Drug: Placebo — Matching placebo, multiple doses
  Arms: Placebo
Drug: RO6811135 — multiple ascending doses
  Arms: RO6811135

SUMMARY:
This randomized, double-blind, placebo-controlled, multiple ascending dose study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of RO6811135 in patients with type 2 diabetes mellitus. Patients will be randomized to receive either RO6811135 or placebo daily for 2 weeks, with a follow-up examination 2 to 3 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 65 years of age, inclusive
* Type 2 diabetes mellitus according to WHO criteria diagnosed for at least 3 months prior to screening
* On stable dose of metformin for at least 2 months prior to screening
* Fasting plasma glucose during the screening period </= 240 mg/dL
* Hemoglobin A1c (HbA1c) levels at screening >/= 6.5% and </= 10.5%
* Evidence of insulin secretory capacity at screening
* Body mass index (BMI) 27 to 42 kg/m2, inclusive
* Females of child-bearing potential and males with female partners of child-bearing potential must agree to use effective contraception as defined by protocol

Exclusion Criteria:

* Type 1 diabetes
* Acquired or secondary forms of diabetes such as those resulting from pancreatic surgery/injury, cystic fibrosis related diabetes
* History of acute metabolic complications such as diabetic ketoacidosis or state of hyperosmolar hyperglycemia
* Evidence or history of clinically significant diabetic complications such as clinically severe diabetic peripheral neuropathy, clinically significant nephropathy as judged by the investigator, or pre-proliferative/proliferative diabetic retinopathy as judged by the investigator
* History of severe symptomatic hypoglycemia (requiring assistances of a third party) within 6 months prior to screening
* History or presence of clinically significant concomitant disease or disorder
* Hemoglobin level below the lower limit of reference range at screening
* Pregnant or lactating women
* History of anaphylaxis or severe systemic hypersensitivity or allergic reactions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 5 months

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | Day 1 and Day 14
Pharmacodynamics of RO681135: Blood analysis | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Chula Vista, California
  - Cincinnati, Ohio